CLINICAL TRIAL: NCT00901628
Title: Efficacy and Safety of Periarticular Multimodal Drug Injections in Total Knee Arthroplasty
Brief Title: Periarticular Multimodal Drug Injections in Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Tae Kyun Kim, Joint reconstruction center, Dept. of orthopaedic surgery, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B-0804/056-021
Record Dates: First submitted 2009-05-13; First posted 2009-05-14 (Estimated); Results first posted 2013-01-25 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2012-12

CONDITIONS: Osteoarthritis, Knee
Keywords: periarticular multimodal drug injection
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Ropivacaine; Morphine; Ketorolac; Epinephrine; Cefuroxime

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Periarticular Injection group (Experimental): Periarticular injection with ropivacaine, morphine, ketorolac, epinephrine, cefuroxime
  Interventions: Drug: ropivacaine; Drug: morphine sulfate; Drug: ketorolac; Drug: epinephrine; Drug: cefuroxime
- No Injection group (No Intervention): usual postoperative care without periarticular injection

INTERVENTIONS:
Drug: ropivacaine — 300mg (0.75%, 40cc) intraoperative periarticular injection
  Arms: Periarticular Injection group
Drug: morphine sulfate — 10mg intraoperative periarticular injection
  Arms: Periarticular Injection group
Drug: ketorolac — 30 mg intraoperative periarticular injection
  Arms: Periarticular Injection group
Drug: epinephrine — 300 microgram (1:1000) intraoperative periarticular injection
  Arms: Periarticular Injection group
Drug: cefuroxime — 750mg intraoperative periarticular injection
  Arms: Periarticular Injection group

SUMMARY:
The purpose of this study is to determine whether periarticular multimodal drug injection (PMDI) would provide additional benefits in patients after total knee arthroplasty (TKA) for whom contemporary pain control protocols using the continuous femoral nerve block, intra-venous patient controlled analgesia (IV-PCA)and preemptive oral medications. We hypothesized that PMDI would reduce pain level and consumption of PCA and acute pain rescuer and would provide better functional recovery and patient satisfaction. We also hypothesized that the incidence of side effects and complications of the PMDI would be similar to the No-PMDI.

DETAILED DESCRIPTION:
The preemptive multimodal approaches are regarded as a current standard pain management protocol. Recently, periarticular multimodal drug injection (PMDI) has been considered to be one of the most effective and important component in multimodal approaches. Because the contemporary pain management protocol using the regional anesthesia, continuous femoral nerve block (FNB) and intravenous patient-controlled analgesia (PCA) has been proved significantly improved analgesic effects itself, little information whether the PMDI would provide additional pain relief under this pain management protocol is available. Also, because the safety of the high dose local anesthetics and narcotics has not been clarified, a selective application should be considered to patients who were expected to show better analgesia if there were certain patient related factors to predict the additional pain relief effect of the PMDI. Thus, this prospective double-blind randomized study was conducted to determine whether PMDI would provide additional benefits in patients after total knee arthroplasty (TKA) for whom contemporary pain control protocols using the continuous femoral nerve block, IV-PCA and preemptive oral medications in terms of pain relief, consumption of PCA and acute pain rescuer, patients satisfaction, functional recovery, side effects and complications.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary osteoarthritis
* Scheduled for elective total knee arthroplasty
* Signed written informed consent
* Spinal anesthesia

Exclusion Criteria:

* Patients refusing consents
* inability to use the outcome assessment tools
* Contraindications to regional anesthesia
* severe cardiovascular disease
* allergy or contraindication to drugs used in this study
* pre-existing neurologic disease including psychiatric disorder
* drug abuser

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2008-04; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tae Kyun Kim, MD, PhD, Principal Investigator — Joint Recontruction Center, Seoul National University Bundang hospital
Locations (1):
- Joint Reconstruction Center, Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 101 patients who were scheduled for unilateral total knee arthroplasty recruitment at Joint Reconstruction Center, Seoul National University Bundang hospital from April 2008 to March 2009 were recruited.
Pre-assignment Details: no participant was excluded before assignment
Groups:
- No Injection Group: usual postoperative care using the continuous femoral nerve block, IV-PCA and preemptive oral medications without periarticular injection
Period: Overall Study
Arm/Group | Periarticular Injection Group | No Injection Group
Started | 49 | 52
Completed | 45 | 42
Not Completed | 4 | 10
Not completed — disconnection of catheter | 4 | 8
Not completed — disconnection of drain | 0 | 1
Not completed — peroneal nerve palsy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Periarticular Injection Group | No Injection Group | Total
Number analyzed (Participants) | 49 | 52 | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 8 | 17
  >=65 years | 40 | 44 | 84
Age Continuous [Mean (Standard Deviation); unit: years] | 70.2 (7.1) | 70.1 (4.9) | 70.1 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 48 | 92
  Male | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 49 | 52 | 101

OUTCOME MEASURES:

1. Primary Outcome: Pain( Visual Analog Scale )
Description: An independent investigator who was blinded to randomization assessed pain level using 0 to 10 visual analog scale (VAS) that ranged from 0 (no pain) to 10 (worst imaginable pain)at the night after operation.
Time Frame: the night after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Periarticular Injection Group | No Injection Group
Number analyzed (Participants) | 49 | 52
units on a scale | 2.3 (3.2) | 6.4 (3.4)

2. Secondary Outcome: Intravenous Patient Controlled Analgesia(PCA) Consumption During 24 Hours After Surgery
Description: Fentanyl based PCA consumption via PCA pump (microgram)
Time Frame: 24 hours postoperative
Measure: Mean (Standard Deviation); unit: microgram
Arm/Group | Periarticular Injection Group | No Injection Group
Number analyzed (Participants) | 49 | 52
microgram | 169.4 (273.9) | 262.3 (200.2)

3. Secondary Outcome: Participant Number of Postoperative Nausea and Vomiting During 24 Hours After Surgery
Description: An independent investigator assessed participant number of postoperative nausea and vomiting during 24 hours after surgery. Nausea was defined as a subjective unpleasant sensation associated with awareness of the urge to vomit; and vomiting, as the forceful expulsion of gastric contents from the mouth.
Time Frame: 24 hours after surgery
Measure: Number; unit: participants
Arm/Group | Periarticular Injection Group | No Injection Group
Number analyzed (Participants) | 49 | 52
participants | 22 | 15

4. Secondary Outcome: the Proportion of Patients Who Were Satisfied With the Pain Management
Time Frame: postoperative 7 day
Measure: Number; unit: participants
Arm/Group | Periarticular Injection Group | No Injection Group
Number analyzed (Participants) | 49 | 52
participants | 38 | 39

5. Secondary Outcome: The Proportion of Patients Who Could Raise Leg With Replaced Knee Extended
Time Frame: 24 hours postoperative
Measure: Number; unit: participants
Arm/Group | Periarticular Injection Group | No Injection Group
Number analyzed (Participants) | 49 | 52
participants | 18 | 6

6. Secondary Outcome: Maximal Flexion Angle Degree on Postoperative 7 Day
Description: An independent investigator measured the maximal flexion angle (degree) of replaced knee with 28 centimeter armed goniometer on postoperative 7 day
Time Frame: postoperative 7 day
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Periarticular Injection Group | No Injection Group
Number analyzed (Participants) | 49 | 52
degree | 92.3 (17.3) | 95.2 (13.7)

ADVERSE EVENTS:
Time Frame: within postoperative 30 days
Arm/Group | Periarticular Injection Group | No Injection Group
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/52
Other Adverse Events (participants affected / at risk) | 0/49 | 0/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Periarticular Injection Group (N=49) | No Injection Group (N=52)
participant number of postoperative wound infection (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) — A blinded investigator evaluated postoperative wound at 1 month after surgery, and assessed incidence of postoperative wound complication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes